CLINICAL TRIAL: NCT06465563
Title: Adebrelimab With or Without SHR-8068 in Combination With Cisplatin Plus Gemcitabine as First-line Treatment in Patients With Advanced Biliary Tract Cancer: A Randomized, Open-label, Multicenter, Phase II Study
Brief Title: Adebrelimab With or Without SHR-8068 in Combination With Cisplatin Plus Gemcitabine as First-line Treatment in Patients With Advanced Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-201-BTC
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-07

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This study is a randomized, open-label, multicenter, Phase II clinical trial aimed at evaluating the efficacy and safety of Adebrelimab in combination with Cisplatin Plus Gemcitabine, with or without SHR-8068, as first-line treatment for advanced biliary tract cancer. The primary endpoint of the study is the Objective Response Rate (ORR), assessed by investigators based on RECISTv1.1 criteria
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: SHR-8068, Adebrelimab, Cisplatin and Gemcitabine (Experimental)
  Interventions: Drug: SHR-8068; Drug: Adebrelimab; Drug: Cisplatin; Drug: Gemcitabine
- Arm B: Adebrelimab, Cisplatin and Gemcitabine (Experimental)
  Interventions: Drug: Adebrelimab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: SHR-8068 — SHR-8068
  Arms: Arm A: SHR-8068, Adebrelimab, Cisplatin and Gemcitabine
Drug: Adebrelimab — Adebrelimab
Drug: Cisplatin — Cisplatin
Drug: Gemcitabine — Gemcitabine

SUMMARY:
This study aims to evaluate the efficacy and safety of SHR-8068 and Adebrelimab in Combination With Cisplatin Plus Gemcitabine(CisGem), compared with Adebrelimab in Combination With CisGem, as first-line treatment in patients with Advanced Biliary Tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old, both male and female;
2. Histologically or cytologically confirmed unresectable locally advanced, or recurrent/metastatic biliary tract adenocarcinoma (including gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma);
3. Has not received prior systemic anti-tumor therapy;
4. At least one measurable lesion based on RECIST v1.1 criteria;
5. ECOG PS score: 0-1 points;
6. Expected survival period ≥ 3 months;
7. Adequate organ function;
8. Must take one medically approved contraceptive measure;
9. Patients voluntarily joined the study and signed informed consent.

Exclusion Criteria:

1. history or concurrently has other solid tumor;
2. Patients with liver tumor burden greater than 50% of total liver volume;
3. History of previous hepatic encephalopathy;
4. Patients with biliary obstruction ， at risk of biliary tract infection;
5. Patients with undergone major surgical treatment within 4 weeks before randomization;
6. Patients with any active, known or suspected autoimmune disorder;
7. Patients with active pulmonary tuberculosis;
8. Patients with known history of HIV or active hepatitis;
9. Untreated central nervous system metastasis;
10. Pleural or peritoneal effusion with clinical symptoms;
11. Patients with poorly controlled cardiac clinical symptoms or disease;
12. Patients with abnormal coagulation function and bleeding tendency;
13. Known allergic reaction to Adalimumab or other monoclonal antibodies, or to the trial drug;
14. Patients with other potential factors that may affect the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From Randomization to the first occurrence of disease progression or initiation of new anti-tumor therapy (up to approximately 14 months)
  ORR is defined as the proportion of participants with Complete Response (CR) or Partial Response (PR), as determined by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate | From Randomization to the first occurrence of disease progression or initiation of new anti-tumor therapy (up to approximately 14 months)] (up to approximately 14 months)
  DCR is defined as the proportion of participants with Complete Response (CR), Partial Response (PR) or Stable Disease (SD), as determined by the investigator according to RECIST v1.1.
Progression-Free-Survival (PFS) | From randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first) (up to approximately 14 months)
  PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first).
Duration of Response (DoR) | From the first occurrence of a confirmed objective response to disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first) (up to approximately 14 months)
  DOR is defined as the time from the first occurrence of a confirmed objective response to disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided